CLINICAL TRIAL: NCT02164318
Title: Effects of Exercise and Improved Nitric Oxide Bioavailability on Arteriovenous Fistula Maturation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00054388; R21DK103082 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (No Intervention): Standard of care
- Handgrip training group (Experimental): Perform isometric handgrip exercises for 15 minutes twice per day for a total of 30 minutes
  Interventions: Other: Handgrip training
- Nitroglycerin ointment group (Experimental): Apply 15mg of nitroglycerin ointment to the back of the hand of the surgical arm nightly
  Interventions: Drug: Nitroglycerin ointment
- Combined handgrip training /Nitroglycerin ointment group (Experimental): Perform isometric handgrip exercises for 15 minutes twice each day for a total of 30 minutes and apply 15mg of nitroglycerin ointment to the back of the hand of the surgical arm nightly
  Interventions: Other: Handgrip training; Drug: Nitroglycerin ointment

INTERVENTIONS:
Other: Handgrip training
  Arms: Combined handgrip training /Nitroglycerin ointment group; Handgrip training group
Drug: Nitroglycerin ointment
  Other Names: Nitropaste
  Arms: Combined handgrip training /Nitroglycerin ointment group; Nitroglycerin ointment group

SUMMARY:
This project will examine if enhancing Nitric Oxide (NO) bioavailability increases the rates of arteriovenous fistula (AVF) maturation in end stage renal disease patients requiring vascular access for hemodialysis. To enhance NO bioavailability the study team will utilize a program of forearm exercise training, application of nitroglycerin ointment or both. Goals of this study are (A) to measure if recruited subjects can tolerate the intervention protocols, and determine if dependent variable measures, including surgery outcome, and measurement of physiologic and biologic markers, can be obtained; (B) To measure subject compliance and adherence rates for each of the intervention arms and testing visits; (C) To examine which intervention or combination of interventions demonstrates the strongest preliminary effects in order to estimate power for a pivotal intent to treat trial; and (D) explore group differences in clinical vascular markers and biologic markers in vein tissue.

DETAILED DESCRIPTION:
This project will examine if enhancing Nitric Oxide (NO) bioavailability increases the rates of arteriovenous fistula (AVF) maturation in end stage renal disease patients requiring vascular access for hemodialysis. To enhance NO bioavailability the study team will utilize a program of forearm exercise training, application of nitroglycerin ointment or both.

Following entry into the study, approximately 4 weeks prior to surgery subjects will undergo a series of non-invasive tests of vascular function in the arm of fistula creation. Following this vascular function testing, subjects will follow the intervention treatment for 4 weeks. After 4 weeks of intervention treatment and prior to surgery, the vascular function analysis will be repeated to determine if the interventions had an effect on arm vascular function. Surgery to create the AVF will follow the second vascular function analysis. A discard sample of the vein used to create the AVF and a blood sample will be collected during surgery to assess potential biologic differences between intervention groups. The interventions will be continued until 4 weeks following surgery. Subjects will be followed to determine if the AVF matured and was successfully used for dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy of at least 6 months
2. Chronic kidney disease with anticipated start of hemodialysis within six months or current hemodialysis dependence.
3. Ability to understand and comply with the requirements of the entire study and communicate with the study team.
4. Written informed consent using a document that has been approved by the Duke Human Institutional Review Board.
5. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative pregnancy test and be willing to use contraception until completion of 8 weeks of intervention. This will include abstinence, barrier methods, hormones, or intra-uterine device.

Exclusion Criteria:

1. Patients currently on medication that is contraindicated with nitropaste, including isosorbide nitrate therapy, nitroglycerin, minoxidil, or PDE inhibitors (i.e. Sildenafil).
2. Patients with a diastolic blood pressure below 65 or a systolic blood pressure below 90.
3. Patients with a history of illicit drug use in the previous 5 years.
4. Patients who would require AVF placement before completion of the initial 4 weeks of intervention therapy
5. Patients who are otherwise are not suitable for 8 weeks of handgrip training or nitropaste therapy.
6. Patients under the 18 of age are not eligible for nitropaste interventions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09-01; Primary Completion 2016-02-18 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Lawson, MD/PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Handgrip Training Group: Perform isometric handgrip exercises for 15 minutes twice per day for a total of 30 minutes
  Handgrip training
- Nitroglycerin Ointment Group: Apply 15mg of nitroglycerin ointment to the back of the hand of the surgical arm nightly
  Nitroglycerin ointment
- Combined Handgrip Training /Nitroglycerin Ointment Group: Perform isometric handgrip exercises for 15 minutes twice each day for a total of 30 minutes and apply 15mg of nitroglycerin ointment to the back of the hand of the surgical arm nightly
  Handgrip training
  Nitroglycerin ointment
Period: Overall Study
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group
Started | 4 | 3 | 1 | 3
Completed | 4 | 2 | 1 | 2
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group | Total
Number analyzed (Participants) | 4 | 3 | 1 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 3 | 8
  >=65 years | 2 | 1 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (13.9) | 51.0 (28.0) | 41 (0) | 53.7 (10.1) | 54.7 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 3
  Male | 2 | 3 | 1 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 2 | 10
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 1 | 3 | 11
Dialysis Status [Count of Participants; unit: Participants] — Indicates if patient had initiated dialysis at time of enrollment
  Participants | 1 | 1 | 1 | 0 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index calculated from weight/height
  kg/m^2 | 33.1 (14.7) | 27.6 (5.8) | 33.1 (0) | 27.2 (8.0) | 30.0 (9.7)
Hypertension Status [Count of Participants; unit: Participants] — Number of participants with diagnosis of hypertension at enrollment
  Participants
    Hypertension: Yes | 4 | 3 | 1 | 3 | 11
    Hypertension: No | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (CAD) Status [Count of Participants; unit: Participants] — Number of participants diagnosed with coronary artery disease at enrollment
  Participants
    CAD: Yes | 0 | 1 | 0 | 1 | 2
    CAD: No | 4 | 2 | 1 | 2 | 9
Diabetes Mellitus (DM) Status [Count of Participants; unit: Participants] — Number of participants diagnosed with Diabetes Mellitus at enrollment
  Participants
    DM: Yes | 2 | 2 | 0 | 1 | 5
    DM: No | 2 | 1 | 1 | 2 | 6
History of thrombotic disorder (TD) [Count of Participants; unit: Participants] — Number of participants with a history of stroke, deep vein thrombosis or pulmonary embolism at time of enrollment
  Participants
    TD: Yes | 0 | 1 | 0 | 2 | 3
    TD: No | 4 | 2 | 1 | 1 | 8
Hyperlipidemia Status [Count of Participants; unit: Participants] — Number of participants with a diagnosis of hyperlipidemia at time of enrollment
  Participants
    Hyperlipidemia: Yes | 2 | 2 | 0 | 2 | 6
    Hyperlipidemia: No | 2 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Mature Arteriovenous Fistula (AVF)
Description: Use of AVF for dialysis for dialysis dependent participants, or fistula deemed mature based on physical exam in predialysis participants (diameter >6 mm, blood flow >600 ml by ultrasound or estimated by physical exam).
Time Frame: 3 month post surgery to create AVF
Population: Two subjects withdrew from this study prior to their AVF surgery, therefore they were not included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group
Number analyzed (Participants) | 4 | 2 | 1 | 2
Participants
  Mature AVF: Predialysis | 2 | 0 | 1 | 0
  Mature AVF: dialysis dependent | 0 | 0 | 0 | 1
  Not Mature AVF: predialysis | 0 | 1 | 0 | 1
  Not Mature AVF: dialysis dependent | 2 | 1 | 0 | 0

2. Secondary Outcome: Count of Participants With a Patent Fistula
Description: Determination that AVF is patent (has blood flow, no occlusion).
Time Frame: 3 months post surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group
Number analyzed (Participants) | 4 | 2 | 1 | 2
Participants
  AVF Patent: Yes | 4 | 2 | 1 | 2
  AVF Patent: No | 0 | 0 | 0 | 0

3. Secondary Outcome: Count of Participants Using Their AVF for Dialysis
Description: Successful use of AVF at 12 months in dialysis dependent patients. Not relevant in participants that are predialysis or that discontinue dialysis prior to AVF use.
Time Frame: 12 months post surgery
Population: Only subjects who were on dialysis at 12 months are included in the analysis. Only 5 participants were on dialysis at this time.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group
Number analyzed (Participants) | 2 | 2 | 0 | 1
Participants
  AVF used for dialysis: Yes | 2 | 2 | 0 | 1
  AVF used for dialysis: No | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events that are reported to the study staff by the subject during the intervention phase of the study where the subject is contacted by staff three times per week will be documented."
Arm/Group | Control Group | Handgrip Training Group | Nitroglycerin Ointment Group | Combined Handgrip Training /Nitroglycerin Ointment Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/1 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 1/1 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=4) | Handgrip Training Group (N=3) | Nitroglycerin Ointment Group (N=1) | Combined Handgrip Training /Nitroglycerin Ointment Group (N=3)
Acute uremia/dialysis initiation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke/Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=4) | Handgrip Training Group (N=3) | Nitroglycerin Ointment Group (N=1) | Combined Handgrip Training /Nitroglycerin Ointment Group (N=3)
Head/arm/shoulder pain/discomfort (Musculoskeletal and connective tissue disorders) | 4 (11) | 2 (9) | 1 (4) | 2 (10)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (2) | 1 (2)
Dizziness/Nausea (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (5)
Vomitting (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hypertension/Bradycardia/Chest Pain (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There are no tests of hypotheses. Rather, the interest of this study is in the assessment of the ability of this design to recruit, retain and conduct the intervention in this sample of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No